CLINICAL TRIAL: NCT06384755
Title: Evaluation of a Norwegian Adaptation of the Honest Open Proud Program for Adults With Psychotic and Bipolar Disorders in an Outpatient Setting
Brief Title: Honest Open Proud for Psychotic and Bipolar Disorder in Norway
Acronym: HOP-NOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Carmen Simonsen, Associate Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 645788; 2022_HE2_409659 (Other Grant/Funding Number: The Dam Foundation); 645788 (Other: Regional Ethics Committee (REK), South-East Norway)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Psychotic Disorders; Bipolar Disorder; Disclosure
Keywords: Honest Open Proud program; Psychotic and Bipolar disorders
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: receives the HOP program consisting of four 2-hour sessions divided between week 1, week 2, week 3 and week 6, in groups of 4-10 participants, using a Norwegian adaptation of HOP workbook. The intervention group also receives treatment as usual, consisting of weekly or monthly appointments with a mental health care professional at an outpatient unit in the public mental health care service. The appointments can involve medication management, psychoeducation, support therapy or psychotherapy.
  Interventions: Behavioral: Honest Open Proud program
- Waiting list control group (No Intervention): Waiting list control group: receives only treatment as usual, consisting of weekly or monthly appointments with a mental health care professional at an outpatient unit in the public mental health care service. The appointments can involve medication management, psychoeducation, support therapy or psychotherapy.
  They are offered the HOP program after the trial.

INTERVENTIONS:
Behavioral: Honest Open Proud program — The HOP program involves peer facilitated sessions, in which different stigma and disclosure related topics are introduced to the group, relevant tasks are completed individually, followed by group or two-and-two discussions related to the following topics: week 1 = pros and cons with disclosure, week 2 = different ways of disclosing, week 3 = formulating individual decisions of disclosure, week 6 = evaluating disclosure or non-disclosure in practice.
  Other Names: Coming Out Proud (COP)
  Arms: Intervention group

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility, acceptability and efficacy of a Norwegian adaptation of the group-based intervention 'Honest Open Proud' among adults with psychotic and bipolar disorders in an outpatient setting.

DETAILED DESCRIPTION:
Because people with mental illness experience both public and personal stigma, which is related to lower levels of recovery and wellbeing, it is common to struggle with decisions regarding potential disclosure of mental health difficulties or diagnoses. There are pros and cons with both disclosure and secrecy. Disclosure can lead to social support, followed by improved mental health and reduced public stigma, but also stigmatization and social exclusion. Secrecy can prevent stigmatization but may also lead to social isolation and thus poorer mental health and increased public stigma. Therefore, people with mental illness need help to make strategic decisions about whether, and if so, to whom, when and how they wish to disclose their mental health problems. As contact with other people with mental health difficulties is crucial to anti-stigma interventions, people with mental illness could benefit from meeting peers, especially as role models. This suggests that peer facilitators could be an important feature in a program aiming to help people with mental illness handle stigma and challenges related to disclosure. The Honest Open Proud (HOP) program was developed for this purpose. Because people with psychotic and bipolar disorders experience particularly high levels of both public and personal stigma, which negatively impacts their recovery rates, they may be especially in need of the HOP program.

The investigators aim to evaluate whether a Norwegian adaptation of the HOP group program, which is facilitated by peers, is feasible and acceptable for people with psychotic and bipolar disorders in an outpatient setting. Moreover, whether it helps them handle stigma and disclosure related decisions.

The investigators propose a pilot randomized controlled trial, comparing an intervention group receiving a 6-week Norwegian adaptation of the HOP program to a waiting list control group. Both groups receive treatment as usual. The main research question is whether this intervention is feasible and acceptable. However, efficacy measures tapping change in stigma and disclosure distress, as well as recovery and wellbeing, from before to after the intervention, were included. The aim is to find what effect sizes can be expected in future larger studies in Norway, rather than to find significant differences in effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed current psychotic (F 20) or bipolar disorder (F 30) according to International Classification of Diseases 10th Revision (ICD-10)
* Age 18 to 65
* Ability to provide written informed consent.
* Fluent in Norwegian (needed for self-report measures)
* Experience difficulties with stigma and disclosure regarding mental illness.

Exclusion Criteria:

* Intellectual disability
* Organic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stigma Stress Scale (Rüsch, Corrigan, Wassel et al., 2009; Rüsch, Corrigan, Powell et al., 2009) | Change from T0 to T1 and T2 (assessed at T0 = week 0; T1 =week 3; T2 = week 6)
  8 items, from 1 (strongly disagree) to 7 (strongly agree)

SECONDARY OUTCOMES:
Disclosure Distress (Rüsch et al., 2014a) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  1 item "In general, how distressed or worried are you in terms of secrecy or disclosure of your mental illness to others?", from 1 (not at all) to 7 (very much)
Warwick and Edinburgh Wellbeing Scale (WEMWBS) (Tennant et al 2007) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  14-items, from 1 (not at all) to 5 (all the time)
Satisfaction with life (Lehman, 1988) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  1 item from Lehmans Quality of Life Scale, from 1 (very dissatisfied) to 7 (very satisfied)
The Questionnaire about the Process of Recovery - 15 (QPR-15) (Niel et al 2007) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  15 items short version, from 0 (strongly disagree) to 4 (strongly agree)
Internalised Stigma of Mental Illness Inventory (ISMI-10) (Boyd, Otilingam, & Deforge, 2014) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  10-item short version, from 1 (strongly disagree ) to 4 (strongly agree )
Patient Health Questionnaire-4 (PHQ-9) (Kroenke et al 2009) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  9 items, 0 (not at all) to 3 (nearly every day)
Generalized Anxiety disorder (GAD-7) (Spitzer et al, 2006) | Change from T0 to T2 (assessed at T0 = week 0; T2 = week 6)
  7 items, from 0 (not at all) to 3 (nearly every day)

OTHER OUTCOMES:
Disclosure | Assessed at T1 and T2 (T1= week 3 and T2 = week 6)
  "Have you disclosed your mental illness the last three (or six) weeks?", YES/NO "How satisfied are you with that?", from 1 (very dissatisfied) to 7 (very satisfied)
Feasibility of HOP program | Tracked during trial and evaluated after completion (T2 = week 6)
  Recruitment rates (numbers of participants in number of weeks) and drop-out rates.
Acceptability of HOP program participants | Assessed after T2 = week 6
  Semi-structured focus-group interview about acceptability with HOP program participants
Acceptability of HOP peer facilitators | Assessed after T2 = week 6
  Semi-structured focus-group interview about acceptability with HOP peer facilitators

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Simonsen, PhD, Principal Investigator — Department of Psychology, University of Oslo
Locations (2):
- Norway (2):
  - Nydalen DPS, Division of Mental Health and Addiction, Oslo University Hospital, Oslo
  - Søndre Oslo DPS, Division of Mental Health and Addiction, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
The study protocol can be shared, but not the the actual data.

REFERENCES:
- See also: Description of the project in Norwegian — https://www.oslo-universitetssykehus.no/avdelinger/klinikk-psykisk-helse-og-avhengighet/forsknings-og-innovasjonsavdelingen-i-pha/regionalt-kompetansesenter-for-tidlig-intervensjon-ved-psykoser/apen-og-varsom-om-psykose-og-bipolar-lidelse-bruker-til-bruker